CLINICAL TRIAL: NCT04410640
Title: Ethical Committee at Researches of Ege University
Brief Title: Surgical Planning With Patient-specific Pancreaticobiliary Disease With 3D Models
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Figen GOVSA, Prof. Dr, Senior investigator, Ege University
Other Study IDs: EGE18-6.134
Record Dates: First submitted 2020-03-12; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Surgical Injury
Keywords: Graduate medical education; Personalized medicine
MeSH Terms: conditions — Intraoperative Complications | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: survey — Members chosen for this study group are general surgery residents. A quintet with stations composed of normal pancreaticobiliary anatomy, common bile duct tumor, stony cholecystitis, pancreatic head cancer and cholelithiasis was assembled for the study. Each station contained CT, 3D-STL images and 1:1 solid models of cases. Each imaging method associated with the scenarios of the quintet is observed by the residents of the study. An explanatory assessment measure is being used as data collection method where the perception of each imaging method is being evaluated based on their effectiveness in problem identification as well as their efficiency in diverse diagnosis and pre-surgery organization. Participants' perception of residency training was evaluated with a multi-entry survey. The focus of the survey, which was applied by our team was by domains, self determined decision-making, diverse diagnosis, academic scholarship, and scientific appraisal.

SUMMARY:
Background: Three-dimensional (3D) printing has been increasingly used in medical applications with the creation of accurate patient-specific 3D printed models in medical imaging data. However, research on 3D printing in pancreaticobiliary disease is limited with lack of studies on validation of model accuracy.

Methods: This is a where general surgery residents, are introduced to 5 distinct hepatopancreatobiliary disease scenarios to generate a perception and required to compare their perception level of these cases with computed tomography (CT), 3D images and 1:1 solid models that the pathology, diverse diagnosis and presurgery diagnosis stages can be investigated.

DETAILED DESCRIPTION:
2.1.Research Design This study group are general surgery residents present in Faculty of Medicine, Ege University (n=19). A quintet with stations composed of normal pancreaticobiliary anatomy, common bile duct tumor, stony cholecystitis, pancreatic head cancer and cholelithiasis is assembled for the study. Each station containes CT, 3D-STL images and 1:1 solid models of cases. Each imaging method (CT, 3D-STL image and 3D solid model) associated with the scenarios of the quintet is created in the residents of the study. An explanatory assessment measure is being used as data collection method where the perception of each imaging method is being investigated based on their effectiveness in problem identification as well as their efficiency in diverse diagnosis and pre-surgery organization.

2.2. Selection of the sample cases The patients are chosen among the CT examinations of the ones who referred to Ege University Faculty of Medicine, Department of General Surgery for diagnose and treatment between 2016 and 2018. CT archives are screened and 5 eligible patients (age: 18-62 year) who required hepatopancreatobiliary surgery were selected. Selection of the cases is based on patients with no previous hepatopancreatobiliary operation, pathology leading to dilated biliary duct, and whose radiological imaging results are suitable for modeling. Virtual modeling of pancreaticobiliary pathways of the cases is performed and clinical histories of each case were created.

2.3. Scenarios As a mutual agreement among the specialists in medical education, general surgery, anatomy and radiology, 5 cases identified, are elected to be samples for pancreaticobiliary surgical processes. Having defined these cases, they are further converted into genuine scenarios fully equipped with a past story, medical analysis results and imaging procedures.

Scenarios for 5 cases:

Case 1. Case with normal extrahepatic biliary tract with pancreas. Case 2. Choledochal tumor leading to advanced dilatation and hydropic gallbladder appearance in extrahepatic biliary tract.

Case 3. Acute cholecystitis characterized with extrahepatic biliary dilatation, hydropic gallbladder, thickness in gallbladder wall and biliary sludge with multiple millimeter-sized stones.

Case 4. Pancreatic head cancer with severe dilatation in the pancreatic canal and extrahepatic biliary tract.

Case 5. Choledocholithiasis characterized with dilatation at the extrahepatic biliary tract and 7 mm diameter stone at the distal end of the common bile duct.

2.4. Image post-processing and segmentation Original CT images in Digital Imaging and Communications in Medicine (DICOM) format are converted to a separate workstation with Analyze 12.0 for post-processing and segmentation. A free 3D slicer (version 4.10.1) is employed in the process of attaining DICOM output from CT and MRI segments of the patients. Special attention is paid to the anatomical structures of the biliary tract including left hepatic duct (LHD), right hepatic duct (RHD), and common hepatic duct (CHD) which are segmented. The surface condition of the model is enhanced by implementing a softening filter to the segmented section output. The output is extracted into STL format to enable 3D printing.

2.5. Creating Life-size Patient-Specific 3D Model 3D printers of Mass Portal Pharaoh xd 20 and Form Labs2 are employed throughout the process of preparing the models for printing.

2.6. Quantitative assessment of model accuracy To ensure the model accuracy, measurements of the anatomical landmarks are performed and compared at three stages of the model production, namely, the original CT images, STL file and 3D model. The internal diameter of four anatomical locations is measured from left to right and from anterior to posterior in the following landmarks: CHD, LHD, RHD and common bile ducts. .

2.7. Workshop We performed a systematic review to evaluate of bile tree modelization and 3D printing, as well as the proof of concept of the benefit of 3D solid model in planning interventions. CT images of a patient diagnosed with dilated extrahepatic ducts are used to create the patient-specific, 1-1 scale 3D pancreaticobiliary models including five scenarios as the normal anatomy, common bile duct tumor, stony cholecystitis, pancreatic head cancer and cholelithiasis. For this purpose, scenarios for each case and a five-station carousel are based on the research. For each station, a period of 5-10 minutes is given.

2.8. Survey Participants' perception of residency training is evaluated with a multi-entry survey. In these scenarios, normal pancreaticobiliary organs and cases leading to extrahepatic biliary tract dilatation such as choledochal tumor, acute stone cholecystitis, pancreatic head tumor and cholelithiasis are discussed. Assessment forms for the normal structure of the cases, differential diagnosis and imaging methods in preoperative planning and the location of the 3D solid model are prepared. The forms are then asked to be filled by the residents to discover their opinions on all models. The evaluaton is done on a scale of 10, where (01-10) defines 0 = very low and 10 = the highest rank.

2.9. Statistical analysis Analysis will be submitted into SPSS 24.0 for statistical evaluation mean ± standard deviation format is employed for continuous variables. Any significant differences in the measurements between the original CT images, 3D-STL images and the 3D model are studied by using Wilcoxon Signed Test. Wilcoxon Signed Ranks Test is used to determine any significant differences in the measurements between the original CT images, 3D-STL images and the 3D model. Statistical relevance is stated as a p value of less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* normal pancreaticobiliary anatomy case
* common bile duct tumor case,
* acute calculous cholecystitis,
* pancreatic head cancer
* cholelithiasis
* general surgery residents present in Faculty of Medicine, Ege University

Exclusion Criteria:

* Hepatic disease
* General surgery experts

Ages: 24 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Members chosen for this study group are general surgery residents present in Faculty of Medicine, Ege University
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
compare the effectiveness of the solid model with CT screen, 3D-Standard Tessellation Language (STL) image and 1:1 scale model | 30 minute
  Our aim is to compare the effectiveness of the solid model with CT screen, 3D-Standard Tessellation Language (STL) image and 1:1 scale model in 5 different hepatopancreatobiliary disease scenarios to general surgery residents in terms of recognizing the pathology, differential diagnosis and preoperative preparation stages.

CONTACTS AND LOCATIONS:
Overall Officials: Muhtar S Ersin, Prof. Dr, Study Chair — Faculty of Medicine, Ege University
Locations (1):
- Ege University, Faculty of Medicine, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Our aim is to compare the effectiveness of the solid model with CTimage, 3Dimage and 3Dmodel in 5 different hepatopancreatobiliary disease scenarios presented to general surgery residents in terms of recognizing the pathology, differential diagnosis and preoperative preparation stages. The focus of the survey applied by our team was on domains, decision-making, diverse diagnosis, scientific appraisal. In these scenarios, normal pancreaticobiliary organs and cases leading to extrahepatic biliary tract dilatation such as choledochal tumor, acute stone cholecystitis, pancreatic head tumor and cholelithiasis were discussed. Perception of the anatomical formation, impact of the procedure to diverse diagnosis, operation arrangement and presurgical preparation assistance are the main criteria in the evaluation of every imaging procedure. Any significant differences in the measurements between the CTimages, 3Dimages and the 3Dmodel were obtained by using Wilcoxon Signed Test.